CLINICAL TRIAL: NCT05400356
Title: Dynamics of Immune Map and Outcomes After On-pump Cardiac Surgery: Protocol for a Prospective Cohort Study
Acronym: DIMOCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Du, 37#,Guoxue Road ,Chengdu, Sichuan Province, China, West China Hospital
Other Study IDs: WCH
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: On-pump Valve Surgery or CABG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Complication group: Postoperative complications are defined as postoperative death, vital organ dysfunction, and mechanical ventilation duration greater than 24 hours.The vital organ dysfunction includes new developed acute kidney injury, long-term low cardiac output, severe liver function injury and neurological function injury.
  The time of occurrence is defined as from the beginning of surgery to 30 days after surgery or to discharge from hospital.
  Interventions: Procedure: On-pump valve surgery or CABG
- Non-complication group: Patients with none of postoperative complications which showed in Complication group.
  The time of occurrence is defined as from the beginning of surgery to 30 days after surgery or to discharge from hospital.
  Interventions: Procedure: On-pump valve surgery or CABG

INTERVENTIONS:
Procedure: On-pump valve surgery or CABG — On-pump valve surgery or coronary arterial bypass grafting

SUMMARY:
Although systemic inflammatory response induced by cardiopulmonary bypass is believed as one of main reasons for these adverse events, the involved mechanism is still unclear.This cohort study would include patients undergoing on-pump valve surgery or CABG. By detecting the changes of immune cell expression profile and inflammatory related substances in blood, the spatiotemporal change curve of immune function of patients is drawn for avoiding or treating adverse events.

ELIGIBILITY:
Inclusion Criteria:

* (1) participants aged over 18 years; (2) Participants who scheduled for valve replacement or valvuloplasty, coronary artery bypass under CPB.

Exclusion Criteria:

* (1) participant with a cognitive or mental disorder who is unable to sign an informed consent form; (2) suffering from basic immune system and blood system diseases; (3) pregnancy; (4) preoperative radiotherapy and chemotherapy; (5) receive immunosuppressive drugs within six months;(6) Expected survival time less than 2 years;(7) participated in other intervention clinical trials within 30 days before operation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from West China Hospital of Sichuan University who would undergo cardiac surgery under CPB between June 2022 and December 2022
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
composite outcome | From the beginning of surgery to 30 days after surgery or to discharge from hospital
  the incidence of vital organ injury, which is defined as a composite measure, including postoperative death, vital organ dysfunction, and mechanical ventilation duration greater than 24 hours. And the vital organ dysfunction includes new kidney injury, long-term low cardiac output, severe liver function injury and neurological function injury.

SECONDARY OUTCOMES:
Infection | From the beginning of surgery to 30 days after surgery or to discharge from hospital]
MACCE | From the beginning of surgery to 30 days after surgery or to discharge from hospital]
  including all-cause mortality, myocardial infarction, severe arrhythmias and stroke
Acute lung injury | From the beginning of surgery to 30 days after surgery or to discharge from hospital]
  Acute onset of bilateral infiltrates on the chest readiograph and hypoxaema(PaO2/Fi O2 ratio <300) in the absence of clincial evidence of left atrial hypertension
Gastrointestinal complications | From the beginning of surgery to 30 days after surgery or to discharge from hospital
  including gastrointestinal bleeding and intestinal ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng Y, Ran Y, Wu J, Yang P, Liao X, Zhang J, Meng W, Gou D, Li L, Du L, Lin J. In vitro Validation of a Novel Disposable Remover to Remove Activated Leukocytes Generated During Cardiopulmonary Bypass: A Pilot Study. J Inflamm Res. 2025 Apr 18;18:5355-5370. doi: 10.2147/JIR.S503575. eCollection 2025. PMID 40270561